CLINICAL TRIAL: NCT06308939
Title: Explore the Efficacy and Safety of Eribulin Combined With Sintilimab in the First-line Treatment of Unresectable Locally Advanced or Metastatic HER2-negative Breast Cancer
Brief Title: Eribulin Combined With Sintilimab as First-line Treatment for Unresectable Locally Advanced or Metastatic HER2-negative Breast Cancer:A Multicenter, Single-arm,Phase II Clinical Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Shao Xiying, Medical team leader, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-198
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; HER2-negative; Eribulin; Sintilimab; First-line Treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eribulin Combined With Sintilimab (Experimental): Eribulin: 1.4mg/m^2 day1、8，repeated every 3 week. Sintilimab: 500mg once every three weeks.
  Interventions: Drug: Eribulin; Drug: Sintilimab

INTERVENTIONS:
Drug: Eribulin — 1.4mg/m^2 day1、8，repeated every 3 week.
  Other Names: eribulin mesylate
Drug: Sintilimab — 500mg once every three weeks.

SUMMARY:
This is a multicenter, single-arm,Phase II clinical trial to explore the efficacy and safety of Eribulin combined with Sintilimab in the first-line treatment of unresectable locally advanced or metastatic HER2-negative breast cancer.

DETAILED DESCRIPTION:
Eribulin: According to the standard dose,1.4mg/m^2 day1、8，repeated every 3 week. After 6 cycles, the investigator decided whether to continue treatment depending on the patient's tolerance.

Sintilimab: 500mg once every three weeks. The patients were treated until disease progression or intolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent. 2. Women aged 18 years or older. 3. Eastern Cooperative Oncology Group(ECOG) has a physical fitness score of 0 or 1. 4. Life expectancy is more than six months. 5. Diagnosed as HER2-negative metastatic breast cancer. 6. There was at least one measurable lesion according to RECIST 1.1. 7.Patients with HR-positive HER2-negative metastatic breast cancer received first-line endocrine therapy, including endocrine therapy alone or in combination with a CDK4/6 inhibitor. 8.In the neoadjuvant or adjuvant stage, patients who had received treatment with anthracyclines or taxanes had recurrence or metastasis more than 6 months after the last administration. 9.Patients who are HR-positive can receive first-line endocrine therapy. 10.Good organ function. 11.Fertile female patients must have a negative serum pregnancy test within seven days prior to study treatment and consent to effective contraceptive use for 180 days from screening to the last dose of study treatment. 12.Female patients must agree not to breastfeed during the study period or for 180 days after the last dose of study therapy.

Exclusion Criteria:

* 1.In the metastatic stage, previous use of Eribulin or immunotherapy or other drug chemotherapy. 2.Patients enrolled in any interventional clinical trial at the same time and received the investigational therapy ≤ four weeks prior to initiation of the regimen or at least five half-lives of the investigational drug. 3.Patients who had received radiation therapy with bone marrow coverage >20% within two weeks before the start of treatment, except for minor palliative radiation therapy more than one week before the first day of the study. 4.Patients with a visceral crisis, and requiring chemotherapy. 5.Patients allergic to Eribulin or Sintilimab. 6.

Patients received blood transfusions ( platelets or red blood cells ) within 4 weeks before the initiation of treatment. 7.Patients received colony stimulating factors ( such as granulocyte colony stimulating factor [ g-CSF ], granulocyte macrophage colony stimulating factor or recombinant erythropoietin ) within 4 weeks before the start of treatment. 8.A history of platelet transfusion for chemotherapy-induced thrombocytopenia or prior cancer treatment (lasting > 4 weeks and associated with recent treatment) is known to result in ≥ grade 3 hematological toxicity. 9.The patient had any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML). 10.Patients have a severe, uncontrolled medical condition, a non-malignant systemic disease, or an active, uncontrolled infection. 11.Patients diagnosed, detected, or treated for another type of cancer within ≤2 years prior to beginning regimen therapy. 12.Patients with brain metastases or pial metastases uncontrolled. 13.Patients have received an allogeneic bone marrow transplant or double umbilical cord blood transplant. 14.Patients cannot swallow oral medications. 15.Patients with gastrointestinal disorders that may interfere with the absorption of investigational drugs. 16.Patients have had systemic active autoimmune disease (i.e., disease modulators, corticosteroids, or immunosuppressants) within the past two years.

17.Patients with a history of human immunodeficiency virus, active-hepatitis -B or C.

18.Pregnant or nursing women. Fertile adults without effective contraceptive methods.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-03-08 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
  ORR is defined as the percentage of patients who achieved a best overall response of Complete Response (CR) or Partial Response (PR), per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions as assessed by the Investigator: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 24 months
  From date of first dose until the date of first documented progression or date of death from any cause, whichever came first.
Clinical Benefit Rate (CBR) | up to 24 months
  Percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD) lasting 24 weeksin the ITT analysis set.
Duration of Overall Response(DoR) | up to 24 months
  ime from first recording to CR or PR to disease progression or all-cause death.
Time to response (TTR) | up to 24 months
  TR defined as the time from the date of the first dose of study treatment to the first objective tumor response when CR or PR is observed.
Overall survival (OS) | up to 24 months
  Time to death from any cause from the date of first dose of study treatment
adverse event(AE) | Throughout the experiment, assessed up to 24 months.
  Evaluation performed using the National Cancer Institute (NCI)- Standard for Common Terminology for Adverse Events (CTCAE)v.5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- zhejiangCH, Hangzhou, Zhejiang, China